CLINICAL TRIAL: NCT04770831
Title: An Observational Study of Patients With Recurrent Progressive or Refractory Neuroblastoma or Malignant Pheochromocytoma or Paraganglioma Who Receive 131 I- MIBG
Brief Title: Patients Who Receive 131 I-MIBG
Status: Withdrawn | Type: Observational
Why Stopped: difficult enrollment, no subjects consented or enrolled
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00081388; 00047671 (Other: Advarra IRB); LCI-PED-NEU-MIBG-001 (Other: Atrium Health)
Record Dates: First submitted 2021-02-16; First posted 2021-02-25 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Brain and Nervous System
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm: QOL following MIBG

SUMMARY:
This study is for patients who have have neuroblastoma, pheochromocytoma, or paraganglioma that has come back (relapsed) after treatment or has not gotten better (refractory) with standard treatment. The purpose of this study is to evaluate quality of life and response rate to 131 I-MIBG treatment.

DETAILED DESCRIPTION:
This is an observational, single institution study designed to determine the benefit of 131I-MIBG therapy in subjects with refractory, relapsed or progressive neuroblastoma, malignant pheochromocytoma or paraganglioma, or other neuroendocrine tumors. Response rate, time to progression, and quality of life changes will be evaluated.

ELIGIBILITY:
Inclusion Criteria

Subject must meet all of the following applicable inclusion criteria to participate in this study:

1. Written informed consent, and assent where applicable, and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age greater than or equal to 1 years and less than or equal to 30 years at the time of therapy.
3. Subject is scheduled to receive 131 I-MIBG therapy.
4. Diagnosis of refractory, progressive or relapsed Neuroblastoma, Malignant Paraganglioma, Malignant Pheochromocytoma or other Neuroendocrine Tumors.
5. As determined by the enrolling physician, ability of the subject and parent/caregiver to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria

Subjects meeting the criteria below may not participate in the study:

1. Prior enrollment on LCI-PED-NEU-MIBG-001 trial.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects with refractory, relapsed or progressive neuroblastoma, malignant pheochromocytoma or paraganglioma, or other neuroendocrine tumors will be recruited at Levine Cancer Institute (LCI), Torrence E. Hemby Jr. Pediatric Hematology & Oncology Center, or Atrium Health Levine Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life | For up to 2 years after treatment with 131 I-MIBG
  To assess health related quality of life prior to, during and after therapy with 131 I-MIBG. For subject's ≥8 years of age, their patient reported Peds QL will be compared to their caregiver's perspective.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From on study date to date of progression or death, for up to 5 years
  To assess progression free survival (PFS) to 131I-MIBG therapy for subjects with refractory, relapsed or progressive neuroblastoma, malignant pheochromocytoma or paraganglioma, or other neuroendocrine tumors.
Disease Control Rate | From on study date to off study date, for up to 5 years
  To evaluate disease control rate to 131I-MIBG treatment in subjects with refractory, relapsed or progressive neuroblastoma or other neuroendocrine tumors (not limited to but including malignant pheochromocytoma or paraganglioma).

CONTACTS AND LOCATIONS:
Overall Officials: Javier Oesterheld, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States